CLINICAL TRIAL: NCT04839484
Title: A Prospective, Randomized, Controlled, Multi-center Study of the Safety and Effectiveness of Lumina™ in the Treatment of Nasolabial Folds
Brief Title: LifeSprout Lumina™ Study in the Treatment of Nasolabial Folds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LifeSprout, Inc. (Industry)
Collaborators: Health Policy Associates (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CT001
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Nasolabial Fold

STUDY DESIGN:
Intervention Model Description: Parallel assignment to product to different sides of face, per randomization code. At 12 months subjects may be retreated only with study product (partial cross over potential)
Who Masked: Outcomes Assessor
Masking Description: A blinded evaluator at each site who does not know what patient was treated with what product (per side) scores the patient. Photographic reviewers are also blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Lumina (Experimental): Lumina Dermal Filler injected into 1 nasolabial fold. Optional Touch-up at 3 week visit with same.
  Interventions: Device: Study Product
- Restylane Defyne (Active Comparator): Restylane Defyne Dermal Filler injected into 1 nasolabial fold. Optional Touch-up at 3 week visit with same.
  Interventions: Device: Active Control

INTERVENTIONS:
Device: Study Product — up to 2cc per injection of filler placed into nasolabial fold.
  Other Names: Lumina
  Arms: Lumina
Device: Active Control — up to 2cc per injection of filler placed into nasolabial fold.
  Other Names: Restylane Defyne
  Arms: Restylane Defyne

SUMMARY:
The study will be a prospective, randomized, split-face, double blind, controlled, clinical trial to evaluate the safety and effectiveness of Lumina™ for the treatment of Nasolabial Folds (NLFs). Subjects will be randomized to receive treatment (Lumina™) in one NLF and control (Restylane® Defyne) in the contra-lateral NLF. 118 subjects will be treated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged at least 22 years.
2. Subject has bilateral moderate or severe (grade 3 or 4) NLFs on the WSRS as scored by a live, masked evaluator.
3. Subject willing to abstain from other facial aesthetic procedures in the NLFs through the 12 month (13 month if retreatment at 12 months) follow-up visit which could interfere with treatment outcomes (e.g. facial fillers, skin laser and radiofrequency therapy such as Thermage, chemical re-surfacing, dermabrasion, Botox injections, aesthetic facial surgery, other facial treatments in the NLFs.
4. Subject understands and accepts the obligation to present for all scheduled follow-up visits and is logistically able to meet all study requirements.
5. Subject with facial hair which may obstruct the assessment of the treatment area, must be agreeable with non-laser removal of facial hair prior to assessment visits.
6. Subject willing to provide written informed consent for their participation in the study.

Exclusion Criteria:

1. Subject is a female of childbearing potential (e.g., not postmenopausal for at least one year or has not had a hysterectomy or tubal ligation) not using medically effective birth control (e.g., hormonal methods in use at least 30 days prior to injection or barrier methods such as condom and spermicide in use at least 14 days prior to injection) or is pregnant, lactating, or plans to become pregnant during the study.
2. Subject has participated in a clinical study in which an investigational device or drug was received in the 30 days prior to screening or plans to enroll in such a study during the course of the current study.
3. Subject is an employee or direct relative of an employee of the investigational site or study sponsor.
4. Subject who has received surgery in the NLFs.
5. Subject has a serious or progressive disease, which, in the investigator's judgment, puts the subject at undue risk (e.g. uncontrolled diabetes, autoimmune disease, cardiac pathologies).
6. Subject has an acute inflammatory process or infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events.
7. Subject has a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.
8. Subject has a history of precancerous lesions/skin malignancies.
9. Subject has had an active skin disease within the past 6 months.
10. Subject has scars, infection, rosacea, herpes, acne, blotches or other pathology in the NLFs.
11. Subject has facial hair covering the nasolabial folds that they are unwilling to remove for study assessments.
12. Subject has a past history of streptococcal disease or an active streptococcus infection.
13. Subject has a past history of allergy or hypersensitivity to gram positive bacterial proteins.
14. Subject is predisposed to keloidosis or hypertrophic scarring.
15. Subject has a known history of hyper- or hypo-pigmentation in the NLFs.
16. Subject with known allergy to poly (ε-caprolactone) microfibers, phosphate buffered saline, polyethylene glycol dithiol (PEG-SH), sodium-hyaluronate of bacterial origin, hyaluronic acid or streptococcal protein.
17. Subject has a known history of multiple allergies, allergic/anaphylactic reactions including hypersensitivity to lidocaine or anesthetics of the amide type.
18. Subject has a known bleeding disorder.
19. Subject has received within the past week or plans to receive up to 1 month after treatment high-dose Vitamin E, aspirin, anti-inflammatories, antiplatelets, thrombolytics or any other medication that could increase the risk of bleeding.
20. Subject has received any medication which, in the judgement of the investigator, may interfere with the study objectives.
21. Subject has received within the past 12 months or plans to receive during the study any injections outside of those in the study protocol including non-permanent fillers (e.g., hyaluronic acid, CaHA) or neurotoxin on the face below the orbital rim (forehead is acceptable).
22. Subject has received at any time or plans to receive during the study a permanent filler (e.g., polylactic acid, PMMA, silicone) on the face.
23. Subject has received within the past 2 weeks or plans to receive during the study dermal resurfacing procedures or non-invasive skin tightening on the face.
24. Subject has received in the past 2 weeks or plans to receive during the study prescription facial wrinkle therapies (RENOVA), topical steroids, skin irritating topical preparations, or self-tanning agents on the face.
25. Subject has a known history of rapid weight loss/gain or plans to begin a weight loss program during the study (5% of body weight).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
primary effectiveness Wrinkle Severity Rating Scale (WSRS) | 6 month
  The mean change from baseline of NLFs in the Lumina™ treatment arm will be compared to that of NLFs in the Restylane® Defyne control arm. (5 point scale with 1 being no visible NLF and 5 being extreme, deep and long NLFs)

SECONDARY OUTCOMES:
WSRS other timepoint | 6 weeks, 3, 9, and 12 months
  Individual endpoints at each timepoint of other than 6 month for mean change from baseline on the WSRS scale, as determined by the live, masked evaluator
WSRS proportions | 6 weeks, 3, 6, 9, and 12 months
  proportion of NLFs in the Lumina™ treatment arm compared to that of NLFs in the Restylane® Defyne control arm with ≥1 point improvement from baseline on the WSRS
Global Aesthetics Improvement Scale (GAIS) - Masked Evaluator | 6 weeks, 3, 6, 9, and 12 months
  Individual endpoints for each rater type, as rated by the live, masked evaluator (5 point scale with 1 being most improvement and 5 being worsened)
GAIS Subject | 6 weeks, 3, 6, 9, and 12 months
  Individual endpoints for each rater type, as rated by the study subject.
GAIS Investigator | 6 weeks, 3, 6, 9, and 12 months
  Individual endpoints for each rater type, as rated by treating investigator
FACE-Q (standardized questionnaire developed by Memorial Sloan Kettering) Appraisal of Nasolabial Folds Questionnaire | 6 weeks, 3, 6, 9, and 12 months
  change from baseline for Lumina™ and Restylane® Defyne on the Subject FACE-Q Appraisal of Nasolabial Folds Questionnaire
Visual Analog Scale (VAS) Pain | injection
  pain assessment in NLFs treated with Lumina™ compared to NLFs treated with Restylane® Defyne at initial injection
WSRS Photographics | 6 weeks, 3, 6, 9, and 12 months
  Individual endpoints at each timepoint of 6 weeks, 3, 6, 9, and 12 months for mean change from baseline on the WSRS scale for NLFs treated with Lumina™ compared to NLFs treated with Restylane® Defyne, as rated by a photographic reviewer.
Proportion WSRS photographic | 6 weeks, 3, 6, 9, and 12 months
  proportion of NLFs in the Lumina™ treatment arm compared to that of NLFs in the Restylane® Defyne control arm with ≥1 point improvement from baseline on the WSRS, as determined by a photographic reviewer

OTHER OUTCOMES:
Safety Endpoint | 13 month
  to assess the rate and severity of adverse events from initial treatment through last study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sashank Reddy, M.D., Study Director — LifeSprout, Inc.
Locations (4):
- UZ Brussels - Brussels University Hosptal, Brussels, Belgium
- FACCIA, Lisbon, Portugal
- United Kingdom (2):
  - British Aesthetics, London
  - PHP Aesthetic-PHP Wellness, London

IPD SHARING:
Plan to Share IPD: No